CLINICAL TRIAL: NCT06085508
Title: Fear of MOVEment After Myocardial Infarction or Atrial Fibrillation - Patient Education Via InterneT- a Pilot Study
Brief Title: Fear of MOVEment After MI and AF - InterneT Patient Education
Acronym: MOVE-IT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Sormland County Council, Sweden (Other); Kalmar County Hospital (Other); Region Östergötland (Other)
Responsible Party: Principal Investigator, Anita Karner, Associate professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FORSS-968769; 2023-01-20 (Other Grant/Funding Number: The focus area E-Health)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Infarction; Atrial Fibrillation; Kinesiophobia
Keywords: Kinesiophobia; Myocardial infarction; Atrial fibrillation; Physical activity; Digital patient education
MeSH Terms: conditions — Myocardial Infarction; Atrial Fibrillation; Kinesiophobia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Digital patient education to reduce kinesiophobia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital patient education to reduce kinesiophobia (Experimental): Intervention: Patients with MI and/or AF and kinesiophobia meet 7 times in a group education via Zoom® video meetings with a tutor (nurse, physiotherapist) for 8 weeks and learn about PA, kinesiophobia, AF and/or CAD.
  Interventions: Behavioral: Digital patient education to reduce kinesiophobia after MI and/or AF

INTERVENTIONS:
Behavioral: Digital patient education to reduce kinesiophobia after MI and/or AF — Group-meetings 7 times via Zoom® video with a tutor (nurse, physiotherapist) and learn about PA, kinesiophobia, AF and/or MI. Scenarios start the problem-based learning process involving recorded lectures, behavioral activation, and exposure to PA. Week1: Programme intro. Formulation of individual goals. Home assignment (HA): Lecture PA after MI/AF. Week 2. Discuss HA. Scenario 1: Why PA after MI/AF? (PBL) Formulate questions*. HA: Answer the questions. Week 3. Follow-up HA. Scenario 2. What is MI/AF.* Week 4. Discuss HA. Scenario 3. Living with MI/AF and kinesiophobia - How to make a change?* HA: Map weekly activities, rate as frightening/non-frightening. List PA and choose one to implement. Use SMART GOALS. Lecture: Kinesiophobia. Week 5. Discuss HA. Scenario 4. How can I reduce my fear for PA.* SMART, the activity. Week 6. Discuss HA. Week 7. Own individual work. HA: Evaluate, revise, and perform activities. Week 8. Follow-up of the activity plan. Summarize the program.

SUMMARY:
The overall aim with the project is to evaluate if a digital patient group-education can reduce kinesiophobia and promote physical activity in patients with myocardial infarction (MI) and/or atrial fibrillation (AF)

Research questions

1. Can a digital patient group-education reduce kinesiophobia and promote PA in patients with MI and/or AF?
2. Is a digital patient group-education feasible based on the patients' experiences?

Intervention: Patients with MI and/or AF and kinesiophobia meet 7 times in a group education via Zoom® video meetings with a tutor (nurse, physiotherapist) for 8 weeks and learn about PA, kinesiophobia, AF and/or CAD. The education involves four real life scenarios as a starting point for the learning process inspired by problem-based learning, live stream/recorded lectures/resource, behavioral activation and exposure to PA in order to reduce kinesiophobia and promote PA.

DETAILED DESCRIPTION:
Patients with myocardial infarction (MI) and/or atrial fibrillation (AF) and kinesiophobia meet 7 times in a group education via Zoom® video meetings with a tutor (nurse, physiotherapist) for 8 weeks and learn about physical activity (PA), kinesiophobia, AF and/or MI. The education involves four real life scenarios as a starting point for the learning process inspired by problem-based learning (PBL) live stream/recorded lectures/resources and exposure to PA to reduce kinesiophobia and promote PA.

Intervention: Digital fear of movement programme:

Week 1: Introduction of programme Aim: Patients reflect on expectations of the program and formulate individual goals. Home assignment: Watch digital lecture about PA after MI/AF and SMART Goals.

Week 2: Start Scenario 1: Why PA after MI/AF? Aim: Patients reflect on pros and cons of PA. Discuss lectures watched. Group thoughts and reflections and formulate questions to be answered next meeting (home assignment).

Week 3: Scenario 2: What is MI/AF. Follow-up scenario 1: How does the knowledge affect me. Aim: To reflect on PA and MI/AF. Start scenario 2: Think free and group thoughts and reflections about PA and formulate questions to be answered next meeting (home assignment).

Week 4: Scenario 3: Living with MI/AF and kinesiophobia - How to make a change? Follow-up scenario 2: How does the knowledge affect me. Aim: to identify and become aware of how thoughts affect PA in his/her life. Start scenario 3: Think free and group thoughts and reflections about living with MI/AF and kinesiophobia - How to make a change and formulate questions to be answered next meeting (home assignment). Home assignment: Map activities in a weekly schedule, rate activities as frightening/non-frightening. Make a list of desirable PA and choose one activity to implement. Use SMART GOALS. Watch digital lecture about: Fear avoidance model.

Week 5: Scenario 4: How can I reduce my fear for PA. Follow-up scenario 3: How does the knowledge affect me. Aim: To implement change. Start scenario 4: Think free and group thoughts and reflections about how can I reduce my fear for PA? SMART, the planned activity Week 6: Follow-up scenario 4. Discuss perception and the performance of the activity. What experiences will I take with me in future activities. Discuss how to continue with the activity plan. Aim: To implement change.

Week 7: Own individual work Use documents to plan desirable activity/ies Aim: To enable change. To become aware of and reflect on how thoughts, moods and fears affect his/her life and performance of PA. Home assignment: Evaluate activity plan and revise and perform desired activities.

Week 8: Follow-up of the activity plan of the program. Summarize and discuss the program. Create a plan for maintenance. Aim: To summarize the program and facilitate maintenance of the changes in PA. Create a checklist for coping with future setbacks, identifying tools perceived as helpful by the participant.

ELIGIBILITY:
Inclusion Criteria:

* patients (n=16 with MI and/or AF with kinesiophobia score of > 37.
* Recruitment: around six months after the heart event (MI and or/AF)

Exclusion Criteria:

* ongoing investigation of coronary artery disease and/or atrial fibrillation or other disease that results in a negative prognosis within 1 year.
* patients who have difficulty participating in and cooperating with other people in groups due to, for example, mental illness, obvious abuse of alcohol or drugs, difficulties communicating or reading the Swedish language,
* or participation in other studies that may affect the results are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are asked to state their gender identity
Enrollment: 14 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | At baseline, after the 8-week programme and 3 months after the programme is completed.
  The Tampa Scale of Kinesiophobia - Swedish version for the heart is a scale which comprises 17 items that assess the subjective rating of kinesiophobia. Each item is rated on a 4-point Likert scale with scoring alternatives ranging from "strongly disagree" to "strongly agree". The total score varies between 17 and 68. A high value indicates a high level of kinesiophobia. A cut-off > 37 is defined as a high level of kinesiophobia.

SECONDARY OUTCOMES:
ActiGraph (accelerometer) | At baseline, after the 8-week programme and 3 months after the programme is completed.
  Patient's objective physical activity during day-time for a week. An accelerometer (Actigraph) will be used to objectively assess physical activity (light (LPA), moderate-to-vigorous (MVPA)) and sedentary behaviour. Outcomes will include daily minutes of physical activity and sedentary behaviour, and the proportion and distribution of time spent in each behaviour.
Physical exercise behaviour | At baseline, after the 8-week programme and 3 months after the programme is completed.
  Stages of exercise behaviour change scale is a single-item five-category scale, based on the 'Stages of Change' model was used to measure the level of exercise behaviour. Respondents will be asked to mark one of five statements that most correctly described their current physical exercise level. Each statement corresponded to one of the five stages: precontemplation, contemplation, preparation, action, and maintenance represented an increased order of exercise behaviour.
Self-efficacy | At baseline, after the 8-week programme and 3 months after the programme is completed.
  General self-efficacy scale is a four-point Likert scale ranging from 'not at all true' (1) to 'exactly true' (4). A higher score indicates a higher GSE, which predicts the ability to cope with daily problems and the ability to adapt after experiencing various stressful life events
Heart focused anxiety | At baseline, after the 8-week programme and 3 months after the programme is completed.
  Cardiac Anxiety scale is a 5-point Likert scale with scores ranging from 0 (never) to 4 (always). A high score indicates a greater number of symptoms, greater frequency, or both.
Self-rated health | At baseline, after the 8-week programme and 3 months after the programme is completed.
  EuroQol-visual analogue scales (EQ-VAS) is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Patients' experiences of the digital programme | After the 8-week programme
  Individual semi- structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kärner Köhler, Ass. prof, Principal Investigator — Linkoping University, Dept of Health, Medicine and Care
Locations (1):
- Anita Kärner Köhler, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Maria Bäck at Sahlgrenska University manage the data collection, analysis of the accelerometers together with Charlotta Lans at Kalmar hospital County.
  The whole research group will take part in analyzing the questionnaires.
  Part of the research group will analyze the transcriptions of the semistructured interviews.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: We plan to have all data collected in February 2024